CLINICAL TRIAL: NCT03830970
Title: Effect of Canned Beans of Multiple Varieties in Daily Amounts of 1 Cup and 1/2 Cup on Serum LDL Cholesterol and Other Cardiovascular Disease Risk Biomarkers in Adults With Elevated LDL Cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Canadian Agricultural Partnership Pulse Science Cluster Program (Unknown); The Bonduelle Company (providing the canned beans) (Unknown)
Responsible Party: Principal Investigator, Alison Duncan, Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: REB-18-10-045
Record Dates: First submitted 2019-02-04; First posted 2019-02-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Hypercholesterolemia; Cardiovascular Diseases
Keywords: Mixed Beans
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 cup of canned beans of multiple varieties (Experimental): Consumption of 1 cup of canned beans of multiple varieties each day for 4 weeks
  Interventions: Dietary Supplement: Canned beans of multiple varieties
- 1/2 cup of canned beans of multiple varieties (Experimental): Consumption of 1/2 cup of canned beans of multiple varieties each day for 4 weeks
  Interventions: Dietary Supplement: Canned beans of multiple varieties
- 1 cup of White rice (Other): Consumption of 1 cup of white rice each day for 4 weeks
  Interventions: Dietary Supplement: White Rice

INTERVENTIONS:
Dietary Supplement: Canned beans of multiple varieties — Daily rotation of different varieties of canned beans including black, navy, pinto, red kidney and white kidney
  Arms: 1 cup of canned beans of multiple varieties; 1/2 cup of canned beans of multiple varieties
Dietary Supplement: White Rice — Minute Rice Long Grain White Rice
  Arms: 1 cup of White rice

SUMMARY:
The Bean Study will examine the effects of consuming two daily amounts of canned beans of multiple varieties on fasting serum cholesterol profile in adults with elevated LDL cholesterol.

DETAILED DESCRIPTION:
The Bean Study (TBS) is a a multi-centre, randomized, crossover design study which will examine the effects of consuming two daily amounts of canned beans of multiple varieties on fasting serum cholesterol profile in adults with elevated LDL cholesterol. Participants will consume daily amounts of 1 cup canned beans, ½ cup of canned beans and 1 cup of white rice for 4 weeks each, separated by minimum 4-week washout periods. At the start and end of each 4-week treatment period, fasting blood samples will be collected and analyzed for lipids, glucose insulin and short chain fatty acids (SCFAs). Fecal samples will also be collected and analyzed for SCFA, bile acids and gut microbiota. Body weight and BMI will be also be measured at the start and end as well as mid-way of each treatment period. Finally 3-day food records will be completed mid-way during each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults (≥18 years)
* BMI 18.5-35 kg/m2
* LDL cholesterol 3.0-5.0 mmol/L

Exclusion Criteria:

* Triglycerides ≥3.0 mmol/L
* Diabetes (fasting blood glucose ≥7.0 mmol/L)
* Blood pressure >140/90 mmHg
* Major medical conditions
* Medical or surgical events requiring hospitalization within the last 3 months
* Medication use that would interfere with the study outcomes (e.g. cholesterol-lowering medications, diabetes-related medications, steroids). All other medications are okay if at a stable (3-month) dose
* Antibiotic use within the last 3 months
* Tobacco product use (>5 times per week)
* Cannabis use during the study
* Probiotic supplement use (could do a 1-month washout before study)
* Dietary fibre supplement use (could do a 1-month washout before study)
* NHPs used for cholesterol lowering or glycemic control. All other NHPs are okay if at a stable (3-month) dose.
* Pulse consumption >4 servings per week
* Food allergy or non-food life-threatening allergy
* Pregnant or breastfeeding
* Alcohol consumption (>14 drinks/week or >4 drinks/sitting)
* Recent or intended significant weight loss or gain (>4 kg in previous 3 months)
* National-level or professional athlete
* Overnight shift worker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Fasting serum LDL cholesterol | 4 weeks (28 days)
  Fasting serum LDL cholesterol will be compared among treatments at study day 29 using ANCOVA and including study day 1 as a covariate

SECONDARY OUTCOMES:
Fasting serum total cholesterol, HDL cholesterol and triglycerides | 4 weeks (28 days)
Fasting serum glucose and insulin and HOMA-IR | 4 weeks (28 days)
  Fasting glucose and insulin
Fasting serum and fecal short chain fatty acids | 4 weeks (28 days)
Fecal bile acids | 4 weeks (28 days)
Gut Microbiota | 4 weeks (28 days)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Human Nutraceutical Research Unit, Guelph, Ontario
  - Glycemic Index Laboratories, Inc, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doma KM, Dolinar KF, Dan Ramdath D, Wolever TMS, Duncan AM. Canned Beans Decrease Serum Total and LDL Cholesterol in Adults with Elevated LDL Cholesterol in a 4-wk Multicenter, Randomized, Crossover Study. J Nutr. 2021 Dec 3;151(12):3701-3709. doi: 10.1093/jn/nxab323. PMID 34642756